CLINICAL TRIAL: NCT04766190
Title: DISCO: A Patient Intervention to Reduce the Financial Burden of Cancer
Acronym: DISCO
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Lauren Hamel (Other)
Responsible Party: Sponsor-Investigator, Lauren Hamel, Principal Investigator, Barbara Ann Karmanos Cancer Institute
Organization: Barbara Ann Karmanos Cancer Institute (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 2020-117; RSG-20-026-01 - CPHPS (Other Grant/Funding Number: American Cancer Society)
Record Dates: First submitted 2021-02-10; First posted 2021-02-23 (Actual); Last update posted 2025-05-25 (Actual); Status verified 2025-05

CONDITIONS: Financial Toxicity; Cancer; Question Prompt List; Breast Cancer; Prostate Cancer
Keywords: Financial Toxicity; Cancer; Treatment cost; Patient-provider communication
MeSH Terms: conditions — Financial Stress; Neoplasms; Breast Neoplasms; Prostatic Neoplasms | interventions — Immunization, Secondary

STUDY DESIGN:
Intervention Model Description: The research tests the effectiveness of an application-based ("app") communication intervention designed to improve the frequency and quality of patient-oncologist treatment cost discussions during clinical interactions, and associated measures.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Group 1: Usual Care (Other): The patient will be asked to arrive 30 minutes early to their next scheduled appointment with their oncologist so they can complete a survey.
  The patient will be video recorded at their appointment. The oncologist has agreed to be video recorded. Immediately after this appointment, the patient will be asked to complete another brief survey that takes about 20 minutes. The questions will ask about how the meeting went. The patient's meeting with the oncologist will not be delayed or changed in any way because of this study.
  Interventions: Behavioral: Group 1: Usual Care
- Group 2: The DISCO App (Other): The patient will be asked to arrive 30 minutes early to their next scheduled appointment with their oncologist so they can complete a survey.
  The patient will be shown an iPad with an "app" while waiting to see their oncologist. The app includes a short video and asks questions about the patient's financial concerns. The app will give the patient a list of questions the patient may want to ask their oncologist during their appointment. The patient will then meet with their oncologist. The meeting with the patient's oncologist will be video recorded. The oncologist has agreed to be video recorded. Immediately after meeting the oncologist, the patient will complete another brief survey. The questions will ask about how the meeting went and what the patient thought of the app. The meeting with the oncologist will not be delayed or changed in any way because of this study.
  Interventions: Behavioral: Group 2: The DISCO App
- Group 3: The DISCO App + Booster (Other): The patient will be asked to arrive 30 minutes early to their next scheduled appointment with their oncologist so they can complete a survey.
  The patient will be shown an iPad with an "app" while waiting to see your oncologist. The app includes a short video and asks questions about your financial concerns. The app will give the patient a list of questions they may want to ask their oncologist during their appointment. The patient will then meet with their oncologist. The meeting with their oncologist will be video recorded. The oncologist has agreed to be video recorded. Immediately after meeting their oncologist, they will complete another brief survey. The questions will ask about how the meeting went and what they thought of the app. The patient's meeting with the oncologist will not be delayed or changed in any way because of this study. Two months after that appointment, the patient will be sent a reminder of the information that was presented on the app.
  Interventions: Behavioral: Group 3: The DISCO App + Booster

INTERVENTIONS:
Behavioral: Group 2: The DISCO App — Patients will receive an individually-tailorable cancer treatment cost education and communication intervention delivered on an iPad just prior to meeting with their oncologist.
  Arms: Group 2: The DISCO App
Behavioral: Group 1: Usual Care — Patients randomized to this arm will receive usual care.
  Arms: Group 1: Usual Care
Behavioral: Group 3: The DISCO App + Booster — Patients will receive an individually-tailorable cancer treatment cost education and communication intervention delivered on an iPad just prior to meeting with their oncologist. Then, 2 months later they will receive an intervention booster in the form of an individually-tailored email to remind patients of the contents of the intervention.
  Arms: Group 3: The DISCO App + Booster

SUMMARY:
The DISCO App is designed to improve, during the interaction, patient active participation and patient-initiated oncologist treatment cost discussions, and, in the short term, patient's treatment cost knowledge, self-efficacy for managing both cost and physician interactions, referrals, perceived financial toxicity (i.e., distress and material hardship); in turn, these will affect longer-term outcomes of financial toxicity and adherence.

DETAILED DESCRIPTION:
This work is based on the core scientific premise - that increasing patient active participation and the frequency and quality of treatment cost discussions will decrease the short- and longer-term burdens of financial toxicity through their influence on self-efficacy for managing treatment cost. The focus is on patient self-efficacy for managing treatment cost because it is expected that improved treatment cost education and patient-oncologist treatment cost discussions prompted by the DISCO App will directly improve the self-efficacy needed for patients to proactively manage treatment costs, thus reducing the material and psychological burden of financial toxicity. The DISCO App is not designed to increase patients' ability to pay or reduce the cost of treatment, but it may benefit patients by increasing: their knowledge of treatment costs, their self-efficacy for managing cost, and the likelihood they receive financial and psychological assistance and support. This research is significant because, if successful, reducing the material and psychological burden of financial toxicity will improve the quality of care and work toward achieving health equity. The DISCO App has already been tested for its feasibility and acceptability. The DISCO App will now be tested for its effectiveness in a diverse population of people with solid tumors treated with IV and oral chemotherapies.

ELIGIBILITY:
Inclusion Criteria:

* Oncologists are eligible if they treat patients with breast, prostate, lung, or colorectal cancers at Karmanos Cancer Institute. Data from oncologists will include their self-report data and video-recorded treatment discussions with participating patients.
* Patients: Must be able to read and write in English; have an email account; and are newly diagnosed with breast, prostate, lung or colorectal cancer (stage I-IV) for which systemic therapy is a likely recommended treatment. Data from patients will include their self-report data, video-recorded treatment discussions with participating oncologists, and medical record data

Exclusion Criteria:

-

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 260 (Estimated)
Dates: Start 2021-02-10 (Actual); Primary Completion 2027-08-31 (Estimated); Study Completion 2028-08-31 (Estimated)

PRIMARY OUTCOMES:
Self-efficacy in patient-physician interactions. An example item from the PEPPI scale: How confident are you in your ability to know what questions to ask your doctor? Data will be aggregated using means and standard deviations. | Immediately after the video-recorded patient-physician interaction
  How efficacious patients feel about communicating with physicians. Scale title: Self-efficacy in patient-physician interactions. Minimum = 1; Maximum = 5; higher is a better outcome.
Self-efficacy in managing treatment costs An example item from adapted scale: I am confident I can pay for the direct costs of my treatment. Data will be aggregated using means and standard deviations. | Immediately after video-recorded patient-physician interaction
  How efficacious patients feel about managing their treatment costs. Scale title: Self-efficacy in managing treatment costs. Minimum = 1; Maximum = 5; higher is a better outcome.
Knowledge of types of treatment cost An example item from the original measure: Cancer treatment may cost me in the following ways? Data will be aggregated using frequency counts. | Immediately after video-recorded patient-physician interaction
  If patients know the types of cost associated with cancer treatment
Perceived financial toxicity; Scale title: Adapted Comprehensive score for financial toxicity (COST) measure. | Immediately after video-recorded patient-physician interaction
  Anticipated financial harm due to treatment cost. Scale title: Adapted Comprehensive score for financial toxicity (COST) measure. Minimum = 0; Maximum = 4; lower is a better outcome.
Perceived presence of treatment cost discussion | Immediately after video-recorded patient-physician interaction
  Patient perception that treatment cost discussed with the physician
Patient self-report of level of satisfaction with any treatment cost discussions with physician assessed via an original scale: satisfaction with any treatment cost discussed with the physician that occurred. | Immediately after video-recorded patient-physician interaction
  Scale title: Satisfaction with any treatment cost discussed with the physician that occurred. Minimum = 1; Maximum = 5; higher is a better outcome.
The observed frequency of a cost discussion assessed via an original coding system. Frequency is assessed as the number of distinct cost discussions that occur in each recorded interaction. Higher is a better outcome. | During the video-recorded patient-physician interaction
  Observation of the frequency of a cost discussion. Minimum = 0; Maximum = undefined.
Patient-Centered Communication scale. The observed quality of patient-physician communication assessed a validated coding system. Minimum = 1; Maximum =5; higher is a better outcome | During the video-recorded patient-physician interaction
  Observation of the quality of patient-physician communication.
Referral to social work/financial navigator | Immediately after video-recorded patient-physician interaction
  If the patient was referred to a social worker or financial navigator. The number of patients who receive a referral to a social worker or a financial navigator.

SECONDARY OUTCOMES:
Self-efficacy in patient-physician interactions. An example item from the PEPPI scale: How confident are you in your ability to know what questions to ask your doctor? Data will be aggregated using means and standard deviations. | 1, 3, 6, and 12 months after video-recorded patient-physician interaction
  How efficacious patients feel about communicating with physicians. Scale title: Self-efficacy in patient-physician interactions. Minimum = 1; Maximum = 5; higher is a better outcome.
Self-efficacy in managing treatment costs | 1, 3, 6, and 12 months after video-recorded patient-physician interaction
  How efficacious patients feel about managing their treatment costs. Scale title: Self-efficacy in managing treatment costs. Minimum = 1; Maximum = 5; higher is a better outcome.
  An example item from the adapted scale: I am confident I can pay for the direct costs of my treatment.
  Data will be aggregated using means and standard deviations.
Financial toxicity | 1, 3, 6, and 12 months after video-recorded patient-physician interaction
  The experience of financial harm due to treatment cost. Rate of patients who indicate they are experiencing financial burden due to cancer treatment costs.
Follow up with social work/financial navigator | 1, 3, 6, and 12 months after video-recorded patient-physician interaction
  If the patient followed up with social work/financial navigator if referred.
  Data will be aggregated using frequency counts.
Treatment adherence An example item from the Medical Outcomes Study General Adherence measure: I had a hard time doing what the doctor suggested I do for treating my cancer. | 1, 3, 6, and 12 months after video-recorded patient-physician interaction
  If the patient adhered to the recommended treatment
Treatment-cost related adherence | 1, 3, 6, and 12 months after video-recorded patient-physician interaction
  If the patient was unable to adhere to treatment due to cost
Clinical appointment adherence. The rate of appointments a patient is scheduled for and attends. | 1, 3, 6, and 12 months after video-recorded patient-physician interaction
  If the patient adhered to clinical appointments

OTHER OUTCOMES:
Assessment of the intervention. | Immediately after video-recorded patient-physician interaction
  Patient perceptions of the intervention's usefulness using an original scale.
  An example item from the original measure: The DISCO App helped me ask my doctor my cost questions. Minimum = 1; Maximum = 5; higher is a better outcome.
Assessment of the intervention booster An example item from the original measure: The reminder email or text message was helpful with my cost questions and concerns. | 1 month after the video-recorded patient-physician interaction
  Patient perceptions of the intervention booster's usefulness
Intervention presence in video-recorded patient-physician interaction | During the video-recorded patient-physician interaction
  If the interaction is visible in the video-recorded patient-physician interaction

CONTACTS AND LOCATIONS:
Overall Officials: Lauren Hamel, PhD, Principal Investigator — Barbara Ann Karmanos Cancer Insitute
Locations (1):
- Barbara Ann Karmanos Cancer Institute, Detroit, Michigan, United States

REFERENCES:
- [Derived] Hamel LM, Dougherty DW, Kim S, Heath EI, Mabunda L, Tadesse E, Hill R, Eggly S. DISCO App: study protocol for a randomized controlled trial to test the effectiveness of a patient intervention to reduce the financial burden of cancer in a diverse patient population. Trials. 2021 Sep 17;22(1):636. doi: 10.1186/s13063-021-05593-y. PMID 34535162